CLINICAL TRIAL: NCT00062608
Title: RCT of Written Self-disclosure for Youth Abdominal Pain
Brief Title: Written Self-disclosure for Youth Abdominal Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RCTYAP (completed)
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Abdominal Pain
Keywords: Abdominal
MeSH Terms: conditions — Abdominal Pain

INTERVENTIONS:
Behavioral: Written self-disclosure

SUMMARY:
The aims are to evaluate: (1) the effectiveness of written self-disclosure (WSD) on health status of youth ages 12-18 with functional recurrent abdominal pain (RAP); (2) whether effectiveness of WSD is similar for younger (12-14) and older (15-18) youth with functional RAP; and (3) the feasibility and acceptability of WSD when extended to the pediatric health care setting.We will implement a randomized, controlled trial (RCT) designed to compare health status in 140 youths (ages 12-18) with functional RAP assigned either to standard medical care (SMC) or WSD provided in the health care setting in addition to SMC. Health status will be measured at Baseline and 3- and 6-months thereafter. Primary measures of health status are symptom severity and episode frequency, consistent with the definition of RAP. Secondary measures of health are functional health, psychological distress, health-related quality of life, and health care utilization. Total use and diagnostic tests will index health care utilization, collected for the 6-mos prior to and following Baseline. Mixed model ANOVA or MANOVA will be used to test directional hypotheses corresponding to the specific aims.

ELIGIBILITY:
* Ages 12-18.
* Diagnosis of RAP by the examining pediatric gastroenterologist using Apley's (1975) criteria: (a) 3 episodes of abdominal pain, (b) severe enough to interrupt activities and occurring, (c) over a period of at least 3 months, (d) without an identifiable organic cause (If an organic cause is identified during participation in protocol, then participant is withdrawn from database prior to analysis).
* Free of a known chronic health condition.
* Physical and mental ability to complete the procedures, as judged by Dr. Madan-Swain.
* Consents to complete the protocol over the next 6 months.
* Parent(s) consents to participate and agrees to support the youth in completing the protocol.
* Access to a phone on the days writing sessions are to be completed at home.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States